CLINICAL TRIAL: NCT01206478
Title: A Phase II, Randomized-Controlled, Multicenter Trial of Amitriptyline for Chronic Oral Food Refusal in Children 9 Months to 8 Years of Age
Brief Title: Trial of Amitriptyline for Chronic Oral Food Refusal in Children 9 Months to 8 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann Davis, PhD, MPH, ABPP (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Ann Davis, PhD, MPH, ABPP, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12261; R21HD066629 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Oral Food Refusal
MeSH Terms: interventions — Amitriptyline; Megestrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amitriptyline plus Megestrol (Experimental): Amitriptyline once daily at bedtime plus megestrol starting at visit 2
  Interventions: Drug: Amitriptyline; Drug: Megestrol
- Placebo plus Megestrol (Active Comparator): Matching placebo once daily at bedtime plus megestrol starting at visit 2
  Interventions: Drug: Placebo; Drug: Megestrol

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline 1 mg/kg once daily at bedtime.
  Arms: Amitriptyline plus Megestrol
Drug: Placebo — Placebo (looks like study drug but has no active ingredients) once daily at bedtime.
  Arms: Placebo plus Megestrol
Drug: Megestrol — At Visit 2, after participating in the study for ten weeks, children will receive a prescription for the appetite stimulant megestrol. The dose each child will receive depends on their age and weight. The dose of megestrol is 6 mg/kg divided into two doses per day.

SUMMARY:
Gastrojejunal (G-J) feeding tubes are placed in infants and children who refuse to eat or are unable to eat enough to have normal growth. Although often intended as temporary short-term solutions to medical complications, feeding tubes can become a permanent method for eating.

While tube feeding routinely saves the lives of children who have long term food refusal, continuation of tube feeding can be hard for patients, caregivers, and families. At the current time there are few treatments for helping children move from tube to oral feeding. Some patients may be treated with the help of inpatient programs such as a combination of medical and behavioral techniques to train children to eat orally. These programs typically require hospital stays of 2-4 months.

By doing the current study the investigators hope to learn if the investigational drug amitriptyline is helpful in moving children from tube to oral feeding, and to look at whether or not the treatment of pain helps with this transition.

DETAILED DESCRIPTION:
This research study involves a study drugs called amitriptyline and megestrol. Amitriptyline might help children who have feeding problems with pain and megestrol is known to increase appetite. Amitriptyline and megestrol are liquid syrups that are given by feeding tube daily.

Amitriptyline has not been approved by the United States Food and Drug Administration (FDA) for the treatment of child with feeding problems. Amitriptyline is an investigational drug that is being studied to find out what the side effects are, and whether or not the product works for child with feeding problems. Amitriptyline is approved by the FDA for the treatment of depression.

Megestrol has not been approved by the United States Food and Drug Administration (FDA) for the treatment of children with feeding problems. Megestrol is an investigational drug that is being studied to find out what the side effects are, and whether or not the product works for children with feeding problems. Megestrol has been approved by the FDA for the treatment of adults. Though megestrol is not FDA approved to treat children with feeding problems, it is often used for this purpose.

Megestrol and Amitriptyline both affect the nerve cells that carry pain sensations to and from the brain. Both drugs reduce the intensity of the pain signals going to the part of the brain that feels pain. Each drug attaches to the nerve cell but at separate spots on the nerve cell so pain can be better managed.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria:

1. Males or females 9 months to 8 years 0 months 0 days of age.
2. Able to obtain parental or legal guardian written informed consent from subjects as applicable by local laws and regulations.
3. Subjects must possess the oral motor skills necessary for eating according to Table 1 in the Appendix.
4. Subjects must possess behavioral skills necessary for mealtime according to Table 2 in the Appendix.
5. Subjects must have a history of chronic oral food refusal (3 months of refusing to eat more than 5% of their caloric intake orally) and be fed >95% of their caloric intake through a gastrostomy tube for 3 months or longer.
6. Subjects will be required to have a body mass index for age/gender of 25% or greater prior to beginning the protocol to ensure that subjects are sufficiently nourished.

Exclusion Criteria

Study enrollment will exclude potential subjects with any of the following conditions or taking any of the following medication:

1. Children on MAO inhibitors or who have thyroid problems will be excluded.
2. Children with diabetes or adrenal insufficiency will be excluded.
3. Children with known heart conduction abnormalities.
4. Children taking tricyclic medications.

Ages: 9 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Davis, Ph.D., MPH, ABPP, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia AM, Beauchamp MT, Patton SR, Edwards S, Dreyer Gillette ML, Davis AM. Family mealtime behaviors in children who are tube fed and preparing to transition to oral eating: A comparison to other pediatric populations. J Health Psychol. 2022 Mar;27(4):1014-1020. doi: 10.1177/1359105320982034. Epub 2020 Dec 18. PMID 33339464
- [Derived] Davis AM, Dean K, Mousa H, Edwards S, Cocjin J, Almadhoun O, He J, Bruce A, Hyman PE. A Randomized Controlled Trial of an Outpatient Protocol for Transitioning Children from Tube to Oral Feeding: No Need for Amitriptyline. J Pediatr. 2016 May;172:136-141.e2. doi: 10.1016/j.jpeds.2016.02.013. Epub 2016 Mar 3. PMID 26947568

RESULTS

PARTICIPANT FLOW:
Groups:
- Amitriptyline, Megestrol: Amitriptyline 1 mg/kg: Amitriptyline 1 mg/kg once daily at bedtime. At Visit 2, after participating in the study for ten weeks, children in both Groups 1 and 2 will receive a prescription for the appetite stimulant megestrol. The dose your child will receive depends on your child's age and weight. The dose of megestrol is 6 mg/kg divided into two doses per day.
- Placebo, Megestrol: Placebo: Placebo (looks like study drug but has no active ingredients) once daily at bedtime.
  At Visit 2, after participating in the study for ten weeks, children in both Groups 1 and 2 will receive a prescription for the appetite stimulant megestrol. The dose your child will receive depends on your child's age and weight. The dose of megestrol is 6 mg/kg divided into two doses per day.
Period: Overall Study
Arm/Group | Amitriptyline, Megestrol | Placebo, Megestrol
Started | 9 | 12
Completed | 7 | 7
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: A total of 21 patients were consented to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline, Megestrol | Placebo, Megestrol | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: age (years)] | 3.54 (2.25) | 3.89 (1.84) | 3.73 (1.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: % Calories Taken Orally
Description: Percent Kilocalories (kcal) Obtained Orally. This measure was obtained using the 24 hour food recall, a standardized five-pass method developed by the US Department of Agriculture for use in national dietary surveillance. This measure has been widely used in several large trials and data suggest it is the most valid and reliable method of dietary assessment for children (20). The data were collected at week 0, week 10, and week 24 using standardized probes by highly trained research staff, and parents were presented with paper food models and measuring devices prior to interviews to reference during the recall. Recalls were analyzed with the Nutritional Data System for Research, version 2005; University of Minnesota, Minneapolis, MN.
Time Frame: baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: change in percent kcal obtained orally
Arm/Group | Amitriptyline, Megestrol | Placebo, Megestrol
Number analyzed (Participants) | 7 | 7
change in percent kcal obtained orally | 68.62 (17.29) | 76.89 (15.68)

2. Secondary Outcome: Change in Non-communicating Children's Pain Checklist - Revised (NCCPC-R) Scores
Description: Non-communicating Children's Pain Checklist - Revised (NCCPC-R) used to measure outcome. The NCCPC-R is a 30 item measure intended to assess pain in children who are unable to speak because of cognitive or physical impairments. There are 7 sub-scales including vocal, social, facial, activity, body/limbs, physiological, and eating/sleeping. Each question has a potential score of 0 to 3. Scores are totaled for each sub-scale. Sub-scale scores are then added together for the Total Score. Total Scores can range from 0 to 90. The higher the score, the higher level of pain indicated by the child. This measure was completed by parents at week 0, week 10, and week 24.
Time Frame: baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline, Megestrol | Placebo, Megestrol
Number analyzed (Participants) | 7 | 7
units on a scale | -2.5 (19.85) | -6.86 (8.65)

ADVERSE EVENTS:
Arm/Group | Amitriptyline, Megestrol | Placebo, Megestrol
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

LIMITATIONS AND CAVEATS:
Major weakness was our small sample size, which was directly due to problems with recruitment, which occurred uniformly across sites. The primary reason for refusal was that parents did not want to be randomly assigned to the amitriptyline/placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No